CLINICAL TRIAL: NCT03161730
Title: Comparison of McGrath Videolaryngoscope, Pentax Airway Scope and Macintosh Laryngoscope in a Normal and Cervical Immobilized Manikin by Novice
Brief Title: Comparison of McGrath Videolaryngoscope, Pentax Airway Scope and Macintosh Laryngoscope in Manikin by Novice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, Jong Yeop Kim, Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: AJIRB-MED-DE4-17-026
Record Dates: First submitted 2017-05-17; First posted 2017-05-22 (Actual); Last update posted 2018-01-10 (Actual); Status verified 2018-01

CONDITIONS: Intubation
Keywords: videolaryngoscope, novice

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- McGrath videolaryngoscopy (Experimental): Participants attempt to perform three intubation using McGrath videolaryngoscope in the manikin with the normal airway and difficult airway scenario, respectively.
  Interventions: Other: McGrath videolaryngoscopy
- Pentax videolaryngoscopy (Experimental): Participants attempt to perform three intubation using Pentax videolaryngoscope in the manikin with the normal airway and difficult airway scenario, respectively.
  Interventions: Other: Pentax videolaryngoscopy
- Macintosh laryngoscopy (Active Comparator): Participants attempt to perform three intubation using Macintosh laryngoscope in the manikin with the normal airway and difficult airway scenario, respectively.
  Interventions: Other: Macintosh laryngoscopy

INTERVENTIONS:
Other: McGrath videolaryngoscopy — Participants perform three intubation attempts using McGrath videolaryngoscope in the normal and cervical immobilized manikin by novice
  Arms: McGrath videolaryngoscopy
Other: Pentax videolaryngoscopy — Participants perform three intubation attempts using Pentax Airway Scope in the normal and cervical immobilized manikin by novice
  Arms: Pentax videolaryngoscopy
Other: Macintosh laryngoscopy — Participants perform three intubation attempts using Macintosh laryngoscope in the normal and cervical immobilized manikin by novice
  Arms: Macintosh laryngoscopy

SUMMARY:
The purpose of this study is to compare the intubation time and success rate between videolaryngoscopes (McGrath MAC videolaryngoscope, Pentax Airway Scope) and Macintosh laryngoscope in tracheal intubation in a normal and cervical immobilized manikin by novice airway managers.

ELIGIBILITY:
Inclusion Criteria:

* nurse without experience in tracheal intubation

Exclusion Criteria:

* refusal to consent

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 35 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2017-12-21 (Actual); Study Completion 2017-12-21 (Actual)

PRIMARY OUTCOMES:
intubation time | within 2 min after insertion of laryngoscope into manikin's mouth
  time the blade passed the manikin's tooth until lung expansion with resuscitation bag

CONTACTS AND LOCATIONS:
Locations (1):
- Jong Yeop Kim, Suwon, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Yi IK, Kwak HJ, Lee KC, Lee JH, Min SK, Kim JY. Comparison of McGrath, Pentax, and Macintosh laryngoscope in normal and cervical immobilized manikin by novices: a randomized crossover trial. Eur J Med Res. 2020 Aug 20;25(1):35. doi: 10.1186/s40001-020-00435-0. PMID 32819444